CLINICAL TRIAL: NCT02139683
Title: High Intensity Focused Ultrasound for the Treatment of Fibroadenomata (HIFU-F)
Brief Title: Feasibility Study Assessing the Treatment of Fibroadenomata With a Circumferential Sonication Treatment With HIFU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Theraclion (Industry)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIFU-F
Record Dates: First submitted 2014-02-05; First posted 2014-05-15 (Estimated); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Breast Fibroadenoma
MeSH Terms: conditions — Fibroadenoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HIFU treatment (Experimental): HIFU treatment in patient diagnosed with fibroadenoma
  Interventions: Device: HIFU treatment

INTERVENTIONS:
Device: HIFU treatment — HIFU treatment in patients with fibroadenoma
  Other Names: Echopulse

SUMMARY:
The purpose of this study is to assess the treatment of fibroadenomata with a circumferential sonification treatment with HIFU..

DETAILED DESCRIPTION:
Primary endpoint: fibroadenomata size reduction post-treatment on ultrasound imaging.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years of age
* Fibroadenomata diagnosed according to local hospital protocol; ultrasound alone on patients <25 and ultrasound plus core-biopsy in patients >25 (Graded B2 or less)
* Visible on ultrasound (Graded U2/U3)
* Definitive diagnosis of fibroadenomata confirmed by the Breast multi-disciplinary team meeting (MDT).

Exclusion Criteria:

* Lesion with atypia or suspicion of phyllodes (Graded B3 or greater)
* Pregnant or lactating women
* History of laser or radiation therapy to the targeted breast

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Changes in size of fibroadenomata as recorded on ultrasound imaging | Month 1, Month 3, Month 12

SECONDARY OUTCOMES:
Adverse Events | Month 1, Month 3, Month 12
Patient recorded outcomes measures | Month 1, Month 3, Month 12
  Patient questionnaires and VAS scales
Mean treatment time | Treatment visit date
Cost-effectiveness | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Douek, MD, Principal Investigator — King's College London
Locations (1):
- Kings College London, Guy's & St Thomas' Hospitals, Department of Research Oncology, London, United Kingdom